CLINICAL TRIAL: NCT00578188
Title: Chlamydia Trachomatis Persistence in the Female Gastrointestinal Tract
Status: Withdrawn | Type: Observational
Why Stopped: Study redesigned and re-submitted to UAMS IRB under different study title and IRB number.
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Amy Scurlock, MD, Arkansas Children's Hospital Research Institute
Other Study IDs: IRB # 43921; ACH GL #039005
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Chlamydia Infection
Keywords: Adolescent Health; Sexually transmitted infection; Women's Health
MeSH Terms: conditions — Chlamydia Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, whole blood, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RP100-400: Subjects with Chlamydia. The control group will also be identified with these numbers.

SUMMARY:
The purpose of this study is to determine if Chlamydial infections persist in the rectum of females who have had a sexually transmitted infection of Chlamydia.

ELIGIBILITY:
Inclusion Criteria:

* 11-19 years old
* Female
* Diagnosis of Chlamydia on enrollment visit
* Invitation to participate control group

Exclusion Criteria:

* Age out of range
* Negative Chlamydia screen (unless qualifies for control group)
* Unable to provide needed samples

Ages: 11 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 11-19 year old females from the Arkansas Children's Hospital Adolescent Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Estimated); Study Completion 2008-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Scurlock, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Chlamydia trachomatis genital infections--United States, 1995. MMWR Morb Mortal Wkly Rep. 1997 Mar 7;46(9):193-8. PMID 9072679
- [Background] Dean D, Suchland RJ, Stamm WE. Evidence for long-term cervical persistence of Chlamydia trachomatis by omp1 genotyping. J Infect Dis. 2000 Sep;182(3):909-16. doi: 10.1086/315778. Epub 2000 Aug 17. PMID 10950788
- [Background] Jones RB, Rabinovitch RA, Katz BP, Batteiger BE, Quinn TS, Terho P, Lapworth MA. Chlamydia trachomatis in the pharynx and rectum of heterosexual patients at risk for genital infection. Ann Intern Med. 1985 Jun;102(6):757-62. doi: 10.7326/0003-4819-102-6-757. PMID 3888022
- [Background] Cotter TW, Ramsey KH, Miranpuri GS, Poulsen CE, Byrne GI. Dissemination of Chlamydia trachomatis chronic genital tract infection in gamma interferon gene knockout mice. Infect Immun. 1997 Jun;65(6):2145-52. doi: 10.1128/iai.65.6.2145-2152.1997. PMID 9169744
- [Background] Igietseme JU, Portis JL, Perry LL. Inflammation and clearance of Chlamydia trachomatis in enteric and nonenteric mucosae. Infect Immun. 2001 Mar;69(3):1832-40. doi: 10.1128/IAI.69.3.1832-1840.2001. PMID 11179361
- See also: Arkansas Children's Hospital Main Page — http://www.archildrens.org